CLINICAL TRIAL: NCT07057141
Title: Effect of Biomimetic Hydroxyapatite-Based Toothpaste and Mouthwash on Dental Sensitivity in Patients With Gingival Recession: A Randomized Controlled Clinical Trial
Brief Title: Biomimetic Hydroxyapatite Toothpaste and Mouthwash for Reducing Dental Sensitivity
Acronym: SENS-BIOREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SENSBIOREPAIR
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Tooth Sensitivity; Gingival Recession Generalized Moderate; Gingival Recession Localized Moderate
Keywords: Dental Hypersensitivity; Tooth Sensitivity; Gingival Recession; Dentin Hypersensitivity; Hydroxyapatite; Biomimetic Hydroxyapatite; Toothpaste; Mouthwash; Visual Analogue Scale (VAS); Shiff Air Index; Desensitizing Agents; Oral Health
MeSH Terms: conditions — Dentin Sensitivity; Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Toothpaste (Active Comparator): 50 participants will receive a single 30-second application of Biorepair Total Protection toothpaste. The intervention aims to reduce dental sensitivity in patients with gingival recession. Clinical indices (Schiff Air Index and VAS) will be assessed before and after application.
  Interventions: Device: Biorepair Total Protection Toothpaste
- Trial Group - Mouthwash (Experimental): 50 participants will receive a single 30-second application of Biorepair high-density mouthwash. The intervention aims to reduce dental sensitivity in patients with gingival recession. Clinical indices (Schiff Air Index and VAS) will be assessed before and after application.
  Interventions: Device: Biorepair High-Density Mouthwash

INTERVENTIONS:
Device: Biorepair Total Protection Toothpaste — Application of Biorepair Total Protection toothpaste for 30 seconds, performed once in a clinical setting. The aim is to reduce dental sensitivity in patients with gingival recession.
  Arms: Control Group - Toothpaste
Device: Biorepair High-Density Mouthwash — Application of Biorepair High-Density mouthwash for 30 seconds, performed once in a clinical setting. The aim is to reduce dental sensitivity in patients with gingival recession.
  Arms: Trial Group - Mouthwash

SUMMARY:
This randomized controlled clinical trial evaluates the effectiveness of a biomimetic hydroxyapatite-based toothpaste and mouthwash in reducing dental sensitivity in patients with gingival recession. A total of 100 participants will be randomly assigned to two groups. The control group will receive Biorepair Total Protection toothpaste, and the trial group will receive Biorepair high-density mouthwash. Both products will be applied for 30 seconds. Dental sensitivity will be assessed before and after treatment using the Shiff Air Index and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 70;
* Subjects with gingival recession and tooth sensitivity;
* Subjects who have agreed to give their free written informed consent to participate in the study.

Exclusion Criteria:

* Male and female subjects who are not adults;
* Subjects without gingival recessions;
* Subjects without dental sensitivity;
* Subjects with poor participation or insufficient motivation to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Dental Sensitivity Measured by the Schiff Air Index | T0 (baseline) and T1 (immediately post-treatment, same visit)
  Variation in dental sensitivity scores assessed using the Schiff Air Index at baseline (T0) and after a 30-second application of either toothpaste or mouthwash (T1). The Schiff scale ranges from 0 (no response) to 3 (painful response to air stimulus), with higher scores indicating greater sensitivity.

SECONDARY OUTCOMES:
Change in Pain Perception Measured by the Visual Analogue Scale (VAS) | T0 (baseline) and T1 (immediately post-treatment, same visit)
  Variation in perceived pain intensity related to dental sensitivity, reported by the patient using the Visual Analogue Scale (VAS) at two timepoints: T0 (baseline) and T1 (immediately after 30-second treatment with either toothpaste or mouthwash). The VAS is a 10 cm horizontal line ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.